CLINICAL TRIAL: NCT07299292
Title: Castration With Abiraterone 250 mg Without LHRH Analogs or Blockers in Patients With Prostate Cancer Requiring Hormonal Intensification (Multicenter Phase 2)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SMED Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TN-2025-0003
Record Dates: First submitted 2025-12-09; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer (Diagnosis)
Keywords: prostate cancer; castration; abiraterone; hormonal intensification
MeSH Terms: conditions — Prostatic Neoplasms; Disease | interventions — abiraterone; Food; Prednisone

STUDY DESIGN:
Intervention Model Description: * Initial Intervention (Day 0-40):
    * Day 0: Testosterone and PSA measurement.
    * Abiraterone acetate 250 mg PO with lunch.
    * Prednisone 5-10 mg/day (either 5 mg/day or 5 mg every 12 h, at investigator's discretion).
    * No ADT until completion of Day 30 evaluation.
  * After Day 30:
    * If the patient achieves castration (primary endpoint met) or not, continue standard indicated treatment (add ADT from Day 31, continue AAP as planned, ± docetaxel/AAP).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single-cohort (Experimental): Abiraterone 250 mg with food + prednisone, without LHRH analogs or blockers (ADT), achieves castration-level testosterone at 30 days in ≥80-90% of cases.
  Interventions: Drug: Abiraterone 250 mg with food + prednisone

INTERVENTIONS:
Drug: Abiraterone 250 mg with food + prednisone — Abiraterone 250 mg with food + prednisone, without LHRH analogs or blockers (ADT), achieves castration-level testosterone at 30 days in ≥80-90% of cases

SUMMARY:
Hypothesis

The use of Abiraterone 250 mg with food + prednisone, without LHRH analogs or blockers (ADT), achieves castration-level testosterone at 30 days in ≥80-90% of cases.

DETAILED DESCRIPTION:
Design

* Type: Phase 2, prospective, open-label, multicenter, single-cohort.
* Inclusion Criteria:

  * Patients with standard indication for intensification:

    * M0 high/very high risk candidates for RT (Abiraterone [ABI] for 2 years + ADT for 3 years per STAMPEDE), or
    * mHSPC: candidates for doublet (ADT+ABI) or triplet (ADT+Docetaxel+ABI); without ADT during the first 30 days.

Objectives and Endpoints

Primary:

1. Proportion of patients with serum testosterone ≤50 ng/dL (and sensitivity analysis ≤20 ng/dL) at Day 30 (±3) without receiving ADT.
2. Time to castration (first day with T ≤50 ng/dL within D1-D30).

Secondary:

* Absolute and % change in PSA between D0 and D30; PSA50 and PSA90 rates at D30.
* Safety (CTCAE v5.0): hypertension, hypokalemia, hepatotoxicity, fluid retention, adrenal insufficiency.

Procedures and Timeline

* Screening (≤7 days): consent, medical history, ECOG, BP, ECG, labs: CBC, liver profile, creatinine, K+, PSA, testosterone.
* Day 0: start ABI 250 mg + prednisone 5-10 mg/day; education on "with food" administration.
* Day 30 (±3): AE, BP, K+, LFT, T, PSA → endpoint evaluation.
* Safety follow-up: until Day 60.

Ethical and Regulatory Considerations

* In Argentina and Bolivia, time to access intensified treatment with Abiraterone (doublet or triplet) exceeds two months in the public system, so waiting time is not altered and patients may benefit from early intensified castration if trial is positive.
* The 250 mg "with food" regimen has pharmacokinetic/economic support in literature; detailed in consent. Multiple studies confirm ABI 250 mg with food equals 1000 mg, and NCCN guidelines recommend this dosing in low-access settings. The SPARE study evaluated safety of ABI without ADT in metastatic castration-resistant prostate cancer, showing equivalence.
* The 30-day window without LHRH is limited, and all patients will receive standard treatment.

Rescue and Safety Criteria • Key AE management:

* Hypokalemia: supplement; consider eplerenone (preferred over spironolactone for lower androgenic interaction); adjust steroid.
* Hypertension: optimize antihypertensives.
* Hepatotoxicity: pauses/adjustments per AAP guidelines.

Sample Size and Justification

* One-sample binomial test to reject p≤0.70 (unacceptable null) in favor of p≥0.90 (target).
* With n=24 per cohort and success defined as ≥20/24 patients achieving castration at D30:

  * α (one-sided) ≈ 0.042 if true p=0.70.
  * Power ≈ 0.91 if true p=0.90.

Variables and Analysis

* Primary: proportion with T ≤50 ng/dL at D30 (main analysis) and T ≤20 ng/dL (sensitivity).

  o Estimate 95% CI and one-sided binomial test vs 70%. Cohort success if ≥20/24 meet criteria.
* Secondary:

  * PSA: absolute and % change, PSA50/PSA90 rates at D30.
  * Safety: AE rates (CTCAE v5.0).

Quality and Logistics

* Testosterone measurement (validated method; preferably LC-MS/MS) to avoid variability.
* Written instructions for administration with food (same time, similar meal).
* Home BP and AE recording (card/app).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Histologically confirmed prostate adenocarcinoma.
* Treated at Hospital Durand (Argentina) or Instituto Oncológico del Oriente Boliviano (Bolivia).
* Indicated for hormonal intensification (high/very high risk candidates for RT, or mHSPC for doublet/triplet).
* No prior ADT.
* ECOG 0-2; adequate hepatic/renal function; K+ ≥3.5 mmol/L; controlled BP.

Exclusion Criteria:

* Hypersensitivity to ABI/prednisone; moderate-severe hepatic impairment; uncontrolled hypertension; refractory hypokalemia.
* Concurrent therapy with strongly contraindicated/inducing drugs affecting ABI levels without possibility of adjustment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Response rate | 3 months
  Response per PCWG3

CONTACTS AND LOCATIONS:
Locations (3):
- Hospital Carlos A Durand, Buenos Aires, Argentina
- Spain (2):
  - Hospital San José, Hermosillo
  - Instituto Oriente Boliviano, Santa Cruz de la Sierra